CLINICAL TRIAL: NCT06569537
Title: Comparison of Compounded Topical Anesthetics for Pain Relief of Intense Pulsed Light, Pulse Dye Laser, and Microneedling Treatments
Brief Title: Comparison of Compounded Topical Anesthetics
Status: Recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Dartmouth-Hitchcock Medical Center (Other)
Responsible Party: Principal Investigator, Brian.J.Simmons, Director of Clinical Trials, Dartmouth-Hitchcock Medical Center
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Supportive Care
Other Study IDs: STUDY02002464
Record Dates: First submitted 2024-08-22; First posted 2024-08-26 (Actual); Last update posted 2025-12-16 (Actual); Status verified 2025-12

CONDITIONS: Procedural Pain
MeSH Terms: conditions — Pain, Procedural | interventions — Lidocaine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Left Side BLT (Experimental): Subjects will receive topical BLT applied to the left side of the face and 4% Lidocaine applied to the right side of the face prior to treatment.
  Interventions: Drug: Lidocaine topical; Drug: BLT
- Left Side Lidocaine (Experimental): Subjects will receive topical 4% Lidocaine applied to the left side of the face and 4% BLT applied to the right side of the face prior to treatment.
  Interventions: Drug: Lidocaine topical; Drug: BLT

INTERVENTIONS:
Drug: Lidocaine topical — 4%
Drug: BLT — Topical Benzocaine 20%/ Lidocaine 8%/Tetracaine 4%

SUMMARY:
The primary objective for this pilot study is to evaluate the efficacy of the compounded topical anesthetic Benzocaine 20%/ Lidocaine 8%/Tetracaine 4% (BLT) compared to 4% Lidocaine topical in providing relief of pain during IPL, PDL, and microneedling procedures.

ELIGIBILITY:
Inclusion Criteria:

* Men and women over 18, but not more than 75 years of age.
* Patients who have a regularly scheduled dermatology appointment for Intense Pulse Light (IPL), Pulse Dye Laser (PDL), or microneedling.

Exclusion Criteria:

* Any subject who has a previous history of allergy, sensitivity, and contraindication to benzocaine, lidocaine, or tetracaine.
* Patients with cardiac/respiratory disease, seizure disorder, or neuropathies.
* Patients who are under treatment for a dermatologic condition that may interfere with the evaluation of the study.
* Pregnant women and women who are breastfeeding.
* Patients who report concurrent use of anxiolytics or opiates, which may interfere with the interpretation of results.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 64 (Estimated)
Dates: Start 2024-10-22 (Actual); Primary Completion 2026-01 (Estimated); Study Completion 2026-01 (Estimated)

PRIMARY OUTCOMES:
Pain as measured by the Numeric Pain Rating Scale (NPRS) | At baseline
  The NPRS pain scale is a segmented numeric version of the visual analog scale (VAS) in which a respondent selects a whole number (0-10 integers) that best reflects the intensity of his/her pain.
Pain as measured by the Wong-Baker Face Pain Rating Scale | At baseline
  This scale shows a series of six faces ranging from a happy face at "no hurt" to a crying face at "hurts worst".

CONTACTS AND LOCATIONS:
Overall Officials: Brian J Simmons, MD, Principal Investigator — Dartmouth Health
Locations (1):
- Dartmouth Hitchcock Dermatology Clinic, Lebanon, New Hampshire, United States

IPD SHARING:
Plan to Share IPD: No